CLINICAL TRIAL: NCT02618187
Title: A Phase 1B Multiple Dose Study to Evaluate the Safety, Tolerability and Microbiome Dynamics of SER-287 in Subjects With Mild-to-Moderate Ulcerative Colitis
Brief Title: A Study to Evaluate the Safety, Tolerability and Microbiome Dynamics of SER-287 in Subjects With Mild-to-Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seres Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SERES-101
Record Dates: First submitted 2015-11-20; First posted 2015-12-01 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Weekly SER-287, after Placebo Pre-Treat. (Experimental): Placebo pre-treatment, followed by once weekly dosing of SER-287 for 8 weeks
  Interventions: Drug: SER-287; Drug: Placebo Pre-Treat
- Daily placebo, after Placebo Pre-Treat. (Placebo Comparator): Placebo pre-treatment, followed by once daily placebo for 8 weeks
  Interventions: Drug: Placebo; Drug: Placebo Pre-Treat
- Daily SER-287, after Vanco. Pre-Treat. (Experimental): Vancomycin pre-treatment, followed by once daily dosing of SER-287 for 8 weeks
  Interventions: Drug: SER-287; Drug: Vancomycin Pre-Treat
- Weekly SER-287, after Vanco. Pre-Treat. (Experimental): Vancomycin pre-treatment, followed by once weekly dosing of SER-287 for 8 weeks
  Interventions: Drug: SER-287; Drug: Vancomycin Pre-Treat

INTERVENTIONS:
Drug: SER-287
  Other Names: Eubacterial Spores, Purified Suspension, Encapsulated
  Arms: Daily SER-287, after Vanco. Pre-Treat.; Weekly SER-287, after Placebo Pre-Treat.; Weekly SER-287, after Vanco. Pre-Treat.
Drug: Placebo
  Arms: Daily placebo, after Placebo Pre-Treat.
Drug: Placebo Pre-Treat
  Arms: Daily placebo, after Placebo Pre-Treat.; Weekly SER-287, after Placebo Pre-Treat.
Drug: Vancomycin Pre-Treat
  Arms: Daily SER-287, after Vanco. Pre-Treat.; Weekly SER-287, after Vanco. Pre-Treat.

SUMMARY:
A Multiple Dose Study to Evaluate the Safety, Tolerability and Microbiome Dynamics of SER-287 in Subjects with Mild-to-Moderate Ulcerative Colitis.

DETAILED DESCRIPTION:
This is a Phase 1b multicenter, randomized, double-blind, placebo-controlled multiple dose study designed to evaluate the safety and tolerability of SER-287, and to evaluate the microbiome alterations and pharmacodynamics associated with two dosing regimens of SER-287 in adult subjects with active mild-to-moderate ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis diagnosed by routine clinical, radiographic, endoscopic and pathologic criteria (preferably confirmed by colonoscopy and pathology records within last 2 years or if unavailable, will need approval by medical monitor) Active mild-moderate UC as determined by sigmoidoscopy within approximately 3 days of randomization to study

Exclusion Criteria:

1. Fever > 38.3°C
2. Known or suspected toxic megacolon and/or known small bowel ileus
3. Known history of Crohn's disease
4. Subjects with serum albumin <2.5 g/dL at baseline
5. CMV polymerase chain reaction (PCR) positive from blood plasma at screening
6. Known stool studies positive for ova and/or parasites or stool culture within the 30 days before enrollment
7. Subjects on cyclosporine or triple immunosuppression, Triple immunosuppression will include any three of the following classes of drugs taken in combination: steroids (i.e., prednisone/budesonide/budesonide MMX), immunosuppressant (i.e., methotrexate/azathioprine/6-mercaptopurine), and/or other immunosuppressant (i.e., tacrolimus, cellcept).
8. Biologic medication (infliximab/ adalimumab/ golimumab/ certolizumab/vedolizumab/ustekinumab/natalizumab) use within 3 months prior to screening
9. Known active malignancy except for basal cell skin cancer, squamous cell skin cancer
10. Subjects with previous colectomy, ostomy, J-pouch, or previous intestinal surgery (excluding cholecystectomy, appendectomy)
11. Subjects with known history of celiac disease or gluten enteropathy
12. Subjects with Clostridium difficile positive stool at Screening Visit
13. Antibiotic use within the prior 1 month before randomization
14. Expected to receive antibiotics within 8 weeks of signing the Informed Consent Form (ICF) (i.e., for planned/anticipated procedure)
15. Received an investigational drug within 1 month before study entry
16. Received an investigational antibody or vaccine within 3 months before study entry
17. Previously enrolled in a SER-109/SER-287 study
18. Received an FMT within the last 6 months
19. Subjects with anatomic or medical contraindications to flexible sigmoidoscopy, including but not necessarily limited to toxic megacolon, gastrointestinal (GI) fistulas, immediate post-operative status from abdominal surgery, severe coagulopathy, large or symptomatic abdominal aortic aneurysm, or any subject where study physician deems subject at significant risk of complications of flexible sigmoidoscopy
20. Unable to stop steroid enemas or suppositories or mesalamine enemas or suppositories before screening visit
21. Unable to stop opiate treatment unless on a stable dose and no increase in dose planned for the duration of the study
22. Unable to stop probiotics before screening visit
23. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy (subjects on maintenance chemotherapy may only be enrolled after consultation with medical monitor)
24. Known allergy or intolerance to oral vancomycin

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Community Clinical Research Network, Marlborough, Massachusetts, United States

REFERENCES:
- [Derived] Henn MR, O'Brien EJ, Diao L, Feagan BG, Sandborn WJ, Huttenhower C, Wortman JR, McGovern BH, Wang-Weigand S, Lichter DI, Chafee M, Ford CB, Bernardo P, Zhao P, Simmons S, Tomlinson AD, Cook DN, Pomerantz RJ, Misra BK, Aunins JG, Trucksis M. A Phase 1b Safety Study of SER-287, a Spore-Based Microbiome Therapeutic, for Active Mild to Moderate Ulcerative Colitis. Gastroenterology. 2021 Jan;160(1):115-127.e30. doi: 10.1053/j.gastro.2020.07.048. Epub 2020 Aug 4. PMID 32763240

RESULTS

PARTICIPANT FLOW:
Groups:
- Weekly SER-287, After Placebo Pre-Treat.: Placebo pre-treatment, followed by once weekly dosing of SER-287 for 8 weeks
  Eubacterial Spores, Purified Suspension, Encapsulated
  Placebo Pre-Treat
- Daily Placebo, After Placebo Pre-Treat.: Placebo pre-treatment, followed by once daily placebo for 8 weeks
  Placebo
  Placebo Pre-Treat
- Daily SER-287, After Vanco. Pre-Treat.: Vancomycin pre-treatment, followed by once daily dosing of SER-287 for 8 weeks
  Eubacterial Spores, Purified Suspension, Encapsulated
  Vancomycin Pre-Treat
- Weekly SER-287, After Vanco. Pre-Treat.: Vancomycin pre-treatment, followed by once weekly dosing of SER-287 for 8 weeks
  Eubacterial Spores, Purified Suspension, Encapsulated
  Vancomycin Pre-Treat
Period: Overall Study
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
Started | 15 | 11 | 15 | 17
Completed (Subjects Completed Visit 12 Endoscopy (8-week treatment)) | 13 | 10 | 13 | 13
Completed (Subjects Completed Visit 13 (short-term safety follow-up)) | 13 | 9 | 11 | 12
Not Completed | 2 | 2 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat. | Total
Number analyzed (Participants) | 15 | 11 | 15 | 17 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (16.12) | 45.8 (15.20) | 47.8 (18.59) | 47.9 (11.18) | 47.1 (15.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 7 | 31
  Male | 6 | 4 | 7 | 10 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 8 | 12 | 15 | 47
  Asian | 0 | 1 | 0 | 1 | 2
  Black or African American | 3 | 1 | 2 | 1 | 7
  Other - Indian | 0 | 1 | 1 | 0 | 2
Montreal Classification [Count of Participants; unit: Participants]
  Ulcerative Proctitis | 0 | 0 | 4 | 2 | 6
  Left-sided UC (distal UC) | 10 | 8 | 5 | 10 | 33
  Extensive UC (pancolitis) | 5 | 3 | 6 | 5 | 19
Severity of UC [Count of Participants; unit: Participants]
  Mild | 6 | 3 | 6 | 10 | 25
  Moderate | 9 | 8 | 9 | 7 | 33
Receiving UC Treatment Prior to or On Date of First Pre-treatment Dose [Count of Participants; unit: Participants]
  No | 2 | 2 | 3 | 6 | 13
  Yes | 13 | 9 | 12 | 11 | 45
Time Since First UC Diagnosis [Mean (Standard Deviation); unit: months] | 149.1 (141.34) | 138.2 (85.91) | 152.9 (143.77) | 142.1 (105.41) | 146.0 (120.12)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of SER-287
Description: Treatment-Emergent Adverse Events Incidence by Treatment, System Organ Class and Preferred Term. The treatment period with SER-287 was eight weeks. All AEs were collected from the date of Informed Consent (up to 17 days of Screening) through Day 92 of the study. All SAEs were collected from the date of Informed Consent through Day 246 of the study.
Time Frame: Day 246
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
Number analyzed (Participants) | 15 | 11 | 15 | 17
Participants
  Gastrointestinal disorders (GI) - total | 7 | 5 | 2 | 8
  GI-Abdominal distension | 0 | 0 | 0 | 1
  GI-Abdominal pain | 3 | 1 | 0 | 4
  GI-Abdominal pain upper | 1 | 0 | 0 | 0
  GI-Abnormal faeces | 0 | 0 | 0 | 1
  GI-Bowel movement irregularity | 0 | 0 | 0 | 2
  GI-Colitis ulcerative (worsening) | 1 | 1 | 0 | 1
  GI-Constipation | 1 | 0 | 2 | 0
  GI-Diarrhoea | 2 | 2 | 0 | 2
  GI-Diarrhoea haemorrhagic | 0 | 1 | 0 | 0
  GI-Dyspepsia | 0 | 1 | 0 | 0
  GI-Faecal incontinence | 0 | 0 | 0 | 1
  GI-Flatulence | 0 | 0 | 0 | 3
  GI-Frequent bowel movements | 1 | 0 | 0 | 0
  GI-Gastrooesophageal reflux disease | 1 | 0 | 0 | 0
  GI-Mucous stools | 0 | 0 | 0 | 1
  GI-Nausea | 3 | 0 | 1 | 1
  GI-Oesophagitis | 0 | 0 | 0 | 1
  GI-Rectal discharge | 1 | 0 | 0 | 0
  GI-Vomiting | 1 | 0 | 0 | 1
  General disorders & administration site conditions | 0 | 1 | 1 | 3
  Immune system disorders | 0 | 0 | 0 | 1
  Infections and infestations | 1 | 3 | 4 | 6
  Injury, poisoning and procedural complications | 0 | 2 | 0 | 0
  Investigations | 0 | 0 | 0 | 1
  Metabolism and nutrition disorders | 0 | 0 | 1 | 1
  Musculoskeletal and connective tissue disorders | 3 | 0 | 2 | 1
  Nervous system disorders | 0 | 0 | 3 | 1
  Psychiatric disorders | 0 | 1 | 1 | 0
  Reproductive system and breast disorders | 0 | 0 | 0 | 1
  Respiratory, thoracic and mediastinal disorders | 1 | 0 | 1 | 2
  Skin and subcutaneous tissue disorders | 0 | 0 | 3 | 1

2. Primary Outcome: Composition of the Intestinal Microbiome
Description: Changes in the composition of the microbiome were characterized by whole metagenomic sequencing (WMS) of subjects' stool samples. Changes in the composition of the microbiome were measured by quantifying the number of unique types of spore-forming bacteria detected in subjects' stool samples after eight weeks of induction treatment versus baseline.
Time Frame: Baseline and 8 weeks
Population: Sensitivity Analysis Population - 1 (all randomized subjects with an evaluable stool sample collected at baseline and one evaluable stool sample collected at Visit 12 or Early Termination (ET) visit collected within a 2 week window surrounding Visit 12)
Measure: Mean (Standard Deviation); unit: Richness of spore-forming species
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
Number analyzed (Participants) | 9 | 6 | 10 | 13
Richness of spore-forming species | 2.333 (8.588) | 0.167 (9.475) | 12.1 (9.871) | 5.615 (9.134)
Statistical Analysis 1: Comparison: Weekly SER-287, After Placebo Pre-Treat. vs Daily Placebo, After Placebo Pre-Treat; Test type: Other — Null hypothesis: the two groups compared show no difference in mean ranks Alternative hypothesis: the two groups compared show a difference in mean ranks; p = 0.766, Wilcoxon (Mann-Whitney); 2-sided
Statistical Analysis 2: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Daily SER-287, After Vanco. Pre-Treat; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.037, Wilcoxon (Mann-Whitney); 2-sided
Statistical Analysis 3: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.313, Wilcoxon (Mann-Whitney); 2-sided
Statistical Analysis 4: Comparison: Weekly SER-287, After Placebo Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.384, Wilcoxon (Mann-Whitney); 2-sided
Statistical Analysis 5: Comparison: Daily SER-287, After Vanco. Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.237, Wilcoxon (Mann-Whitney); 2-sided

3. Primary Outcome: Engraftment of SER-287 Bacteria in All Treatment Arms
Description: The stool microbiomes of SERES-101 subjects, before and after treatment with SER-287, were characterized using whole metagenomic sequencing (WMS). SER-287 drug product was also characterized using WMS. Microbiome engraftment was assessed by the number of spore-forming species in the drug product lots that were also detected in subjects' post-treatment fecal samples but not detected at baseline.
Time Frame: Baseline and 8 weeks
Population: Sensitivity Analysis Population - 1 (all randomized subjects with an evaluable stool sample collected at baseline and one evaluable stool sample collected at Visit 12 or Early Termination (ET) visit collected within a two-week window surrounding Visit 12)
Measure: Mean (Standard Deviation); unit: Richness SER-287 spore-forming species
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
Number analyzed (Participants) | 9 | 6 | 10 | 13
Richness SER-287 spore-forming species | 7.222 (5.974) | 4.333 (1.862) | 16.7 (7.469) | 13.615 (6.225)
Statistical Analysis 1: Comparison: Weekly SER-287, After Placebo Pre-Treat. vs Daily Placebo, After Placebo Pre-Treat; Test type: Superiority — Weekly SER-287, after Placebo Pre-Treat. tested against Daily placebo, after Placebo Pre-Treat., for superiority; p = 0.257, Wilcoxon (Mann-Whitney); 1-sided
Statistical Analysis 2: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Daily SER-287, After Vanco. Pre-Treat; Test type: Superiority — Daily SER-287, After Vanco. Pre-Treat. tested against Daily Placebo, After Placebo Pre-Treat., for superiority; p = 0.001, Wilcoxon (Mann-Whitney); 1-sided
Statistical Analysis 3: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Superiority — Weekly SER-287, After Vanco. Pre-Treat. tested against Daily Placebo, After Placebo Pre-Treat., for superiority; p = 0.001, Wilcoxon (Mann-Whitney); 1-sided
Statistical Analysis 4: Comparison: Weekly SER-287, After Placebo Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Superiority — Weekly SER-287, After Vanco. Pre-Treat. tested against Weekly SER-287, After Placebo Pre-Treat., for superiority; p = 0.009, Wilcoxon (Mann-Whitney); 1-sided
Statistical Analysis 5: Comparison: Daily SER-287, After Vanco. Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Superiority — Daily SER-287, After Vanco. Pre-Treat., tested against Weekly SER-287, After Vanco. Pre-Treat., for superiority; p = 0.168, Wilcoxon (Mann-Whitney); 1-sided

4. Secondary Outcome: Clinical Remission
Description: Defined as a Total Modified Mayo Score <= 2 and an endoscopic subscore <= 1.
  The Total Modified Mayo Score is a measure of UC disease activity which ranges from 0 to 12 points and consists of four subscores (stool frequency, rectal bleeding, endoscopy, and physician global assessment), each graded from 0 to 3, with higher scores indicating more severe disease. The four components are summed together for a composite score, with a higher overall score indicating more severe disease (0 = no disease; 12 = worst disease). The Modified Mayo endoscopic subscore excludes friability from an endoscopic subscore of 1.
Time Frame: 8 weeks
Population: ITT, where the following were counted as missing: missing post-treatment endoscopy; adding UC medication for a flare during the treatment period; early termination prior to Day 48
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
Number analyzed (Participants) | 15 | 11 | 15 | 17
Participants | 2 | 0 | 6 | 3
Statistical Analysis 1: Comparison: Weekly SER-287, After Placebo Pre-Treat. vs Daily Placebo, After Placebo Pre-Treat; Test type: Superiority; p = 0.4923, Fisher Exact; Rate difference (SER-287 - placebo) = 13.3, 95% CI 2-sided [-3.87 to 30.54]
Statistical Analysis 2: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Daily SER-287, After Vanco. Pre-Treat; Test type: Superiority; p = 0.0237, Fisher Exact; Rate difference (SER-287 - placebo) = 40.0, 95% CI 2-sided [15.21 to 64.79]
Statistical Analysis 3: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Superiority; p = 0.2579, Fisher Exact; Rate difference (SER-287 - placebo) = 17.6, 95% CI 2-sided [-0.47 to 35.77]

5. Secondary Outcome: Endoscopic Improvement
Description: Defined as a decrease in endoscopic subscore >= 1
Time Frame: 8 weeks
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
Number analyzed (Participants) | 15 | 11 | 15 | 17
Participants | 5 | 1 | 6 | 4
Statistical Analysis 1: Comparison: Weekly SER-287, After Placebo Pre-Treat. vs Daily Placebo, After Placebo Pre-Treat; Test type: Superiority; p = 0.1973, Fisher Exact; Rate difference (SER-287 - placebo) = 24.2, 95% CI 2-sided [-5.04 to 53.53]
Statistical Analysis 2: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Daily SER-287, After Vanco. Pre-Treat; Test type: Superiority; p = 0.1783, Fisher Exact; Rate difference (SER-287 - placebo) = 30.9, 95% CI 2-sided [0.86 to 60.96]
Statistical Analysis 3: Comparison: Daily Placebo, After Placebo Pre-Treat. vs Weekly SER-287, After Vanco. Pre-Treat; Test type: Superiority; p = 0.6195, Fisher Exact; Rate difference (SER-287 - placebo) = 14.4, 95% CI 2-sided [-11.93 to 40.81]

ADVERSE EVENTS:
Time Frame: Day 246
Description: All AEs were collected from the date of Informed Consent (up to 17 days of Screening) through Day 92 of the study. All SAEs were collected from the date of Informed Consent through Day 246 of the study.
Arm/Group | Weekly SER-287, After Placebo Pre-Treat. | Daily Placebo, After Placebo Pre-Treat. | Daily SER-287, After Vanco. Pre-Treat. | Weekly SER-287, After Vanco. Pre-Treat.
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/11 | 0/15 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11 | 1/15 | 0/17
Other Adverse Events (participants affected / at risk) | 8/15 | 2/11 | 5/15 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weekly SER-287, After Placebo Pre-Treat. (N=15) | Daily Placebo, After Placebo Pre-Treat. (N=11) | Daily SER-287, After Vanco. Pre-Treat. (N=15) | Weekly SER-287, After Vanco. Pre-Treat. (N=17)
Worsening depression (Psychiatric disorders) | 0 | 0 | 1 | 0 — The one case of worsening depression was reported as moderate severity, and probably not or likely not related to study drug, as determined by the investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weekly SER-287, After Placebo Pre-Treat. (N=15) | Daily Placebo, After Placebo Pre-Treat. (N=11) | Daily SER-287, After Vanco. Pre-Treat. (N=15) | Weekly SER-287, After Vanco. Pre-Treat. (N=17)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 4 (5) — Treatment-emergent adverse event
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) — Treatment-emergent adverse event
Diarrhea (Gastrointestinal disorders) | 2 (3) | 2 (3) | 0 (0) | 2 (2) — Treatment-emergent adverse event
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) — Treatment-emergent adverse event
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (2) | 1 (1) — Treatment-emergent adverse event
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) — Treatment-emergent adverse event
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (2) — Treatment-emergent adverse event
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1) — Treatment-emergent adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications must be submitted to Sponsor for review at least 30 days prior to publication. Sponsor can require removal of confidential information other than study data and Site/Investigator agree to consider Sponsor's suggestions with respect to the presentation of study data. Sponsor can force publication to be deferred for a period of up to 60 days in order to file any patents.

DOCUMENTS (3):
  • Study Protocol (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT02618187/Prot_000.pdf
  • Statistical Analysis Plan: SERES-101 SAP (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT02618187/SAP_001.pdf
  • Statistical Analysis Plan: SERES-101 Microbiome SAP (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/87/NCT02618187/SAP_002.pdf